CLINICAL TRIAL: NCT07165834
Title: Take Your Sexuality Back - a Feasibility Study of a New Intervention for Sexually Traumatized Women
Brief Title: Voices of Transformation: A Deep Dive Into the Struggles and Successes of Reclaiming Sexuality After Sexual Trauma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: University of Agder (Other); NTNU Health (sponsor) (Unknown)
Responsible Party: Principal Investigator, Idun Røseth, PhD, Sykehuset Telemark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 829297
Record Dates: First submitted 2025-08-21; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Sexual Abuse; Posttraumatic Stress Symptom; Sexual Trauma
MeSH Terms: conditions — Sexual Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group. "Take your sexuality back" (Experimental): "Take your sexuality back" is a 12 week group intervention for sexually traumatized women.
  Interventions: Behavioral: Treatment group. "Take your sexuality back"

INTERVENTIONS:
Behavioral: Treatment group. "Take your sexuality back" — The intervention is trauma-sensitive and focus both on traumatized sexuality and positive sexuality. It incorporates regulatory skills to prevent re-traumatization when addressing sex-positive themes, thus accommodating a wide range of trauma-related symptoms, sexual shame, sexual dysfunctions, and regulation difficulties. The intervention integrates psychoeducation, exercises, reflections and sharing.

SUMMARY:
This study aims to gain insight into the experiences of participants in the "Take Your Sexuality Back" intervention groups, evaluate the intervention's acceptability, and identify necessary modifications. This study is part of a larger project that seeks to establish a scientific basis for this innovative, group-based treatment to help women who have experienced sexual trauma heal their sexuality. Before implementing the intervention in the healthcare system and initiating a larger randomized controlled trial, the investigators will evaluate the intervention's feasibility and potential efficacy, as well as gain a more comprehensive understanding of treatment outcomes. In addition to collecting quantitative data, it is crucial to gather qualitative data on participants' experiences. In this study, data will be obtained through in-depth interviews with group participants after they complete the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. A history of sexual trauma
2. Experience trauma-related sexual problems
3. Age between 18 and 65 years
4. Enough competence in Norwegian to participate in a psychoeducational group.

Exclusion Criteria:

1. Acute suicidality
2. Serious substance abuse interfering with treatment
3. Severe dissociative or psychotic disorders
4. Current life crisis interfering with treatment
5. Living in an abusive relationship. -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
What are the participants lived experiences of participating in the group intervention "Take your sexuality back" | 1-2 weeks after end of treatment
  In-depth interviews investigating participants experiences and perceptions of the intervention, and how they react to any positive or negative impacts attributed to it. Interviews will be analyzed through a descriptive phenomenological method.

CONTACTS AND LOCATIONS:
Overall Officials: Hege Kersten, PhD, Study Director — Research and Innovation Manager
Locations (1):
- Sykehuset Telemark HF, Skien, Norway

IPD SHARING:
Plan to Share IPD: No
Qualitative data are sensitive and participant anonymity cannot be guaranteed.